CLINICAL TRIAL: NCT04259996
Title: Impact of Serum Progesterone Concentration on the Day of Embryo Transfer in Modified Natural Cycles and Stimulated Cycles on Ongoing Pregnancy Rate
Brief Title: Impact of Serum Progesterone in Modified Natural Cycles and Stimulated Cycles on Ongoing Pregnancy Rate
Acronym: CORPUS-LUTEUM
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1907-VLC-075-EL
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Infertility, Female
Keywords: Progesterone in luteal phase; modified natural cycle; stimulated cycle; clinical pregnancy rate; live birth rate
MeSH Terms: conditions — Infertility, Female | interventions — Progesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MODIFIED NATURAL CYCLE: The term 'modified natural cycle' refers to a natural cycle in which ovulation is triggered by exogenous hCG administration in order to provide optimal timing scheduling embryo transfer. In contrast to the natural cycle, the applied hCG may lead to a different luteal phase profile. Luteal phase support is common clinical practice in those cycles.
  On the day of embryo transfer (ET), eligible patients being transferred one or two good quality embryos on day 5 of development according to the Spanish ASEBIR classification will be informed about the nature of the study, read the informed consent (IC) form and decide if entering into the study. After signing the IC form, a blood test will be performed in a time frame between 1 and 2 hours before the ET.
  The only intervention will be a single determination of serum P and E2 levels immediately before the embryo transfer.
  Interventions: Procedure: PROGESTERONE AND ESTRADIOL SERUM CONCENTRATION MEASUREMENT
- STIMULATED CYCLE: On the day of embryo transfer (ET), eligible patients being transferred one or two good quality embryos on day 5 of development according to the Spanish ASEBIR classification will be informed about the nature of the study, read the informed consent (IC) form and decide if entering into the study. After signing the IC form, a blood test will be performed in a time frame between 1 and 2 hours before the ET.
  The only intervention will be a single determination of serum P and E2 levels immediately before the embryo transfer.
  Interventions: Procedure: PROGESTERONE AND ESTRADIOL SERUM CONCENTRATION MEASUREMENT

INTERVENTIONS:
Procedure: PROGESTERONE AND ESTRADIOL SERUM CONCENTRATION MEASUREMENT — The only intervention will be a single determination of serum P and E2 levels immediately before the embryo transfer.

SUMMARY:
Prospective cohort unicentric study including infertile patients undergoing an embryo transfer in the context of natural or stimulated cycles and receiving luteal phase support with vaginal natural progesterone following the clinical practice in our clinic in IVIRMA Valencia, Spain.

DETAILED DESCRIPTION:
Progesterone as a promoter of endometrial maturation is essential for the process of embryo implantation. The transformation of the endometrium from a proliferative state to a receptive state depends on the adequate progesterone exposure of the endometrium. Therefore, in any assisted reproduction technique (ART) the management of the luteal phase with exogenous administered progesterone, aiming to achieve a receptive endometrial state, is an essential part of the therapy. This important part of infertility-treatment is called luteal phase support (LPS).

Currently, there is a scientific debate and research regarding the timing, the dose and route of administration of exogenous progesterone in ART cycles. For years, the administration of progesterone was based on a "one fits all"- concept, mainly driven from the doctors and patients' preference regarding dose, timing and route of administration of the exogenous progesterone. Due to the lack of solid and evidence-based knowledge, the LPS improving investigating LPS is of outmost importance.

Therefore, improving the LPS is continuously in the focus of research and investigation. Main objectives of those efforts are to clarify the optimal timing, dosage and route of administration of progesterone for every possible ART procedure, in order to improve therapy outcomes. Of special interest in this wide field is the management of LPS in embryo-transfer-cycles such as substituted cycles and modified natural cycles for frozen-thawed cycles, and in fresh embryo-transfers after stimulated cycles.

Measuring serum progesterone levels in the luteal phase of a transfer cycle seems to be a promising approach in resolving the former mentioned doubts. Now, research focuses on luteal-phase serum progesterone levels as a predictor of outcomes. The discovery of certain thresholds of progesterone levels in the serum would give us a handy tool for individualizing the LPS with the main objective to improve outcomes.

Previous studies could show that there exist certain thresholds of serum progesterone in substituted cycles that could be used as a predictor. Furthermore, the same group could show that modifying the dose and the route of administration in the sense of individualizing LPS can improve outcomes.

Considering those results, it remains to clarify if there also exist thresholds of serum progesterone in modified natural cycles and stimulated cycles and if it's possible to improve the results through individualization of LPS the same way as it has been shown for substituted cycles.

The intention of the present study is to carry out the determination of serum progesterone on the day of the embryo transfer to all those patients who are going to be subjected in IVIRMA Valencia to an embryo transfer in a modified natural cycle or a stimulated cycle.

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent prior to any study related procedures
* Women ≤50 years old
* BMI ≤ 40 kg/m2
* Adequate endometrial thickness (>6.5mm) and pattern (Triple A structure) in the proliferative phase
* Regular menstrual cycles

Exclusion Criteria:

* Uterine Pathology, adnexal pathology
* Systemic diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All infertile patients undergoing a fresh or frozen blastocyst transfer (two blastocysts transferred as maximum) from own or donated oocytes; in the context of a modified natural cycle (group A) or a stimulated cycle (group B). As usually performed in our daily clinical practice, all patients will receive hCG to trigger ovulation and maintain the corpus luteum to produce endogenous progesterone. Luteal phase support will be given as usual according to the routine in our center.
Sampling Method: Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 months
  Presence or absence of ongoing pregnancy

SECONDARY OUTCOMES:
Implantation rate | 12 months
  Presence or absence of implantation
Live Birth | 12 months
  Presence or absence of Live Birth
Pregnancy Loss | 12 months
  Presence or absence of pregnancy loss

CONTACTS AND LOCATIONS:
Overall Officials: Elena Labarta, MD, Principal Investigator — IVIRMA VALENCIA
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No